CLINICAL TRIAL: NCT00258908
Title: Immunogenicity and Safety of ADACEL™ (TdcP Vaccine) as Fifth Dose in Children 6-8 Years of Age.
Brief Title: Immunogenicity and Safety of ADACEL™ as Fifth Dose in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TD521
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Results first posted 2009-06-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: ADACEL™; Tetanus; Diphteria; Acellular pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Diphteria, tetanus, and Acellular Pertussis vaccine — 0.5 mL, Intramuscular
  Other Names: ADACEL™

SUMMARY:
To assess the immunogenicity profile of ADACEL™, Tetanus and Diphtheria Toxoids Adsorbed combined with Component Pertussis Vaccine (TdcP Vaccine) one month after administration.

To describe the safety profile of ADACEL™ (TdcP Vaccine) when given as a fifth dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 6 to 8 years on the day of inclusion
* Informed consent form (ICF) signed by parent(s)/legal representative
* Able to attend all scheduled visits and to comply with all trial procedures
* Written documentation of complete primary series and fourth dose of Diphtheria, Tetanus toxoids and whole cell Pertussis vaccine (DTP)
* Parent(s)/legal representative present or fully completed pre-inclusion medical questionnaire

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances with specific focus on subjects who had, after previous administration of DTP or diphtheria and tetanus toxoids and acellular pertussis (DTaP) vaccine, one of the following adverse events

  1. encephalopathy not attributable to another identifiable cause within 7 days of administration of a previous dose
  2. temperature of > 40.5 °C within 48 hours not due to another identifiable cause
  3. collapse or shock-like state (hypotonic-hyporesponsive episode) within 48 hours
  4. persistent, inconsolable crying lasting > 3 hours, occurring within 48 hours
  5. seizure with or without fever occurring within 3 days
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past 3 months
* Any vaccination in the 4 weeks preceding the trial vaccination (except Oral Poliomyelitis Vaccine [OPV])
* Any vaccination planned during the present trial period (except OPV)
* History of diphtheria and/or tetanus and/or pertussis infection (confirmed either clinically, serologically or microbiologically)
* Previous fifth vaccination against diphtheria and/or tetanus and/or pertussis infection with the trial vaccine or another vaccine
* Clinical or serological evidence of systemic illness including Hepatitis B, C or Human Immunodeficiency Virus (HIV)
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures
* Febrile illness (axillary temperature ≥ 37.4 °C) or acute illness on the day of inclusion

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 01 November through 07 December 2005 in 1 medical clinic in Taiwan
Pre-assignment Details: A total of 115 participants that met the inclusion and exclusion criteria were recruited for the study; 112 were vaccinated and included in the final analysis and this report.
Groups:
- ADACEL™ Group: Participants received 1 dose of ADACEL™ (TdcP vaccine)
Period: Overall Study
Arm/Group | ADACEL™ Group
Started | 112 (3 participants were not vaccinated and were not included in the final analysis and in this report.)
Completed | 112
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ADACEL™ Group
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 112
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (0.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 55
Region of Enrollment [Number; unit: participants]
  Taiwan | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody (Anti-diphtheria, Anti-tetanus, and Anti-pertussis Toxoids) Responses Pre- and Post-vaccination
Description: Immunogenicity profile of ADACEL™ (TdcP vaccine) antibody (anti-diphtheria, anti-tetanus, and anti-pertussis) responses at Day 0 and Day 28 Post-vaccination.
Time Frame: Day 0 and Day 28 Post-vaccination
Population: Seroprotection to each vaccine antigen was evaluated in the per-protocol immunogenicity population
Measure: Number; unit: Percentage of participants
Arm/Group | ADACEL™ Group
Number analyzed (Participants) | 112
Percentage of participants
  Anti-diphtheria (≥ 0.01 IU/mL, Day 0) | 95
  Anti-diphtheria (≥ 0.01 IU/mL, Day 28) | 99
  Anti-diphtheria (≥ 0.1 IU/mL, Day 0) | 55
  Anti-diphtheria (≥ 0.1 IU/mL, Day 28) | 99
  Anti-tetanus (≥ 0.01 IU/mL, Day 0) | 100
  Anti-tetanus (≥ 0.01 IU/mL, Day 28) | 100
  Anti-tetanus (≥ 0.1 IU/mL, Day 0) | 90
  Anti-tetanus (≥ 0.1 IU/mL, Day 28) | 100
  Anti-pertussis toxoid (≥4-fold rise, Day 28) | 88
  Anti-Filamentous Haemagglutinin ≥4-fold rise Day28 | 88
  Anti-Fimbriae Types 2 & 3 (≥4-fold rise, Day 28) | 87
  Anti-Pertactin (≥4-fold rise, Day 28) | 99

2. Primary Outcome: Geometric Mean Titers (GMTs) of Anti-diphtheria, Anti-tetanus, and Anti-pertussis Toxoids Pre- and Post-vaccination
Description: GMTs and 95% confidence intervals of anti-diphtheria, anti-tetanus, and anti-pertussis toxoids responses at Day 0 and Day 28 Post-vaccination.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Geometric Mean Titers were evaluated in the per-protocol immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ADACEL™ Group
Number analyzed (Participants) | 112
Titers
  Anti-diphtheria - Day 0 | 0.120 [0.093 to 0.156]
  Anti-diphtheria - Day 28 | 4.87 [3.67 to 6.47]
  Anti-tetanus - Day 0 | 0.386 [0.311 to 0.479]
  Anti-tetanus - Day 28 | 18.8 [15.9 to 22.2]
  Anti-pertussis toxoid - Day 0 | 9.5 [7.53 to 12.0]
  Anti-pertussis toxoid - Day 28 | 189 [147 to 243]
  Anti-Filamentous Haemagglutinin - Day 0 | 16.7 [13.1 to 21.4]
  Anti-Filamentous Haemagglutinin - Day 28 | 234 [203 to 269]
  Anti-Fimbriae Types 2 and 3 - Day 0 | 31.2 [24.8 to 39.1]
  Anti-Fimbriae Types 2 and 3 - Day 28 | 940 [697 to 1268]
  Anti-Pertactin - Day 0 | 8.89 [7.02 to 11.3]
  Anti-Pertactin - Day 28 | 312 [251 to 388]

3. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site and Systemic Reactions Post-vaccination
Description: The percentage of participants reporting solicited injection site and systemic reactions within 8 days after vaccination with ADACEL™ (TdcP vaccine) when given as a fifth dose
Time Frame: Within 8 days of vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | ADACEL™ Group
Number analyzed (Participants) | 112
Percentage of Participants
  Any solicited injection site reaction | 67
  Any Injection site pain | 59
  Gd3 Injection site pain(inj limb movement reduced) | 4
  Any Injection site erythema | 33
  Grade 3 Injection site erythema (≥ 5 cm) | 6
  Any Injection site swelling | 37
  Grade 3 Injection site swelling (≥ 5 cm) | 5
  Any solicited systemic reaction | 58
  Any Fever | 10
  Grade 3 Fever (≥ 39.0 °C) | 0
  Any Headache | 17
  Grade 3 Headache (prevents daily activities) | 1
  Any Malaise | 31
  Grade 3 Malaise (prevents daily activities) | 0
  Any Myalgia | 53
  Grade 3 Myalgia (prevents daily activities) | 1

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from day of vaccination to 28 days post-vaccination.
Arm/Group | ADACEL™ Group
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 10/112
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL™ Group (N=112)
Nasopharyngitis (Infections and infestations) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.